CLINICAL TRIAL: NCT02996123
Title: Biting Force in Heat Cured Acrylic Resin Versus CAD/CAM Maxillary Single Denture Bases: A Randomized Controlled Trial .
Brief Title: Biting Force in Heat Cured Acrylic Resin Versus CAD/CAM Maxillary Single Denture Bases
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Erfan Gamal El Dein, Dr, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EKF 54324
Record Dates: First submitted 2016-12-12; First posted 2016-12-19 (Estimated); Last update posted 2016-12-19 (Estimated); Status verified 2016-12

CONDITIONS: Bites, Human
MeSH Terms: conditions — Bites, Human

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- cad/cam maxillary dentures (Experimental): single maxillary dentures fabricated by cad/cam method
  Interventions: Other: cad/cam maxillary dentures
- conventional dentures (Active Comparator): heat cured single maxillary dentures
  Interventions: Other: cad/cam maxillary dentures

INTERVENTIONS:
Other: cad/cam maxillary dentures — patients wearing cad/cam designed and milled dentures

SUMMARY:
measuring difference in biting force between (computer aided design/computer aided manufacturing) maxillary dentures and conventional ones.

DETAILED DESCRIPTION:
measuring difference in biting force using i-load device with followup period of 6 months

ELIGIBILITY:
Inclusion Criteria:

1. Patients with completely edentulous maxillary ridge with minimum undercuts, opposing a partially edentulous ridge.
2. Mean age of 50-75 years of age.
3. The edentulous ridges should be covered by firm healthy mucosa.
4. Systemically free; no history of diabetes, chemotherapy, and radiotherapy.
5. Co-operative patients.

Exclusion Criteria:

1. Patients with severely resorbed maxillary ridge
2. Previous history of radiotherapy or chemotherapy.
3. Patients with xerostomia
4. Patients with neuromuscular and hormonal disorders
5. Patients with severe bony or soft tissue undercuts
6. Patients with large tongue
7. Patients with limited mouth opening
8. Patients with known history of allergy, especially to acrylic resin

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-11 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Biting Force in Heat Cured acrylic resin versus CAD/CAM Maxillary Single Denture Bases | 6 month

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo university, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
charts with measurements and readings collected will be recorded and available